CLINICAL TRIAL: NCT00002375
Title: A Multicenter, 24-Week Study of the Safety, Pharmacokinetics, and Activity of the Coadministration of Indinavir and Nelfinavir in HIV-1 Seropositive Patients
Brief Title: Safety and Effectiveness of Giving Indinavir and Nelfinavir to HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 246H; MK-0639; 061-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nelfinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to treat HIV-infected patients with indinavir (IDV) plus nelfinavir (NFV), 2 anti-HIV medications.

It is thought that IDV plus NFV will be a safe drug combination for treating HIV.

DETAILED DESCRIPTION:
It is hypothesized that the administration of indinavir with nelfinavir will be generally safe and well tolerated.

This is a parallel, time-lagged, 2-stage, multiple-dose, 24-week study in HIV-1 seropositive patients. In the 3-week, randomized, double-blind phase of Stage A, patients receive either indinavir plus nelfinavir (Group A1: 9 patients) or indinavir placebo plus nelfinavir placebo (Group A2: 3 patients) for the first week. In Week 2, patients in Group A1 have the nelfinavir dose increased. This dose escalation for nelfinavir is contingent upon the patient having completed 1 week of the study drugs without experiencing Grade 3 or worse toxicity and/or serious drug-related adverse events. Patients in Group A2 continue to receive placebo until Week 3, at which time they receive indinavir plus nelfinavir (initial dose), while patients in Group A1 continue with indinavir plus nelfinavir (escalated dose). At Week 4 all patients in Stage A (including those originally assigned to receive placebo) receive open-label indinavir plus nelfinavir (escalated dose) for the remainder of the 24 weeks.

After at least 6 patients in Stage A have completed at least 2 weeks of therapy with nelfinavir plus indinavir with acceptable tolerability, Stage B begins. In the 2-week, randomized, double-blind phase of Stage B, patients receive either indinavir plus nelfinavir (Group B1: 9 patients) or indinavir placebo plus nelfinavir placebo (Group B2, 3 patients). After 2 weeks, all patients in Stage B (including those originally assigned to receive placebo) receive open-label indinavir plus nelfinavir for the remainder of the 24 weeks.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count of at least 100 cells/mm3.
* Have a plasma viral load (level of HIV in the blood) of at least 30,000 copies/ml.
* Are at least 18 years old.

Exclusion Criteria

You will not be eligible for this study if you:

* Have ever been treated with any protease inhibitors (PIs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Treatment Ctr / Dept of Medicine and Pediatrics, San Diego, California
  - Univ of Pittsburgh / Graduate School of Public Health, Pittsburgh, Pennsylvania